CLINICAL TRIAL: NCT01115387
Title: Genetics of Age Related Maculopathy
Brief Title: GARM II: A Study on the Genetics of Age-related Maculopathy
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Jules Stein Eye Institute (Other); University of Pittsburgh (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Michael B. Gorin, Professor of Ophthalmology, University of California, Los Angeles
Other Study IDs: 08-11-008; 5R01EY009859 (NIH)
Record Dates: First submitted 2010-04-26; First posted 2010-05-04 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Age-related Macular Degeneration; Age-related Maculopathy
Keywords: Age-related macular degeneration; AMD; Genetic risk; Environmental risk factors; Complex genetic disorder; Age-related maculopathy; Risk modeling; Smoking; Light exposure; Sleep apnea; Fundus Photography; Macula; Drusen; Wet AMD; Dry AMD; Geographic atrophy; Vitamins & supplements
MeSH Terms: conditions — Macular Degeneration; Smoking; Sleep Apnea Syndromes; Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ARM at risk individuals: A group of 1,500 participants (from 49 to 65 years old) who have at least one parent with age related maculopathy.
  These individuals with ARM-affected parents and relatives have a substantially higher risk (6-12 fold) of developing ARM than the general population. They will be followed prospectively with fundus photography every two years and questionnaires (distributed over six month intervals) to assess external risks for ARM development in order to investigate genotype-phenotype correlations of early onset clinical features of ARM.
  Interventions: Other: Observational-1
- Partners/Spouses of ARM at risk individuals: A group of 1,500 participants (from 49 to 65 years old) who are the spouses/partners of individuals with ARM affected parents.
  We will invite the partners or spouses to participate in order to compare their risk of developing ARM with those individuals with an increased risk of ARM based on a positive family history.
  Interventions: Other: Observational-1
- ARM affected individuals and relatives.: Individuals who have experienced vision loss from ARM and have at least one brother or sister who also has experienced vision loss from ARM can participate in the study. They also need to have at least one adult child (from 49 to 65 years old) who wishes to participate in this study.
  We will allow for additional recruitment to compensate for additional family members (such as parents, aunts and uncles) who wish to participate as well as to address potential drop out and those who may be deemed ineligible based on review of their medical and/or eye records. As many as 4000 individuals in this group will be allowed to enroll.
  Interventions: Other: Observational-2

INTERVENTIONS:
Other: Observational-1 — Multiple questionnaires detailing family history, medical history, visual symptoms, smoking, environmental and dietary exposures.
  Prospective photography of the retina to detect early ARM-related changes A saliva or blood sample for genetic testing.
  Groups: ARM at risk individuals; Partners/Spouses of ARM at risk individuals
Other: Observational-2 — A limited number of questionnaires and prior clinical documentation from eye care professionals of eye status with respect to ARM.
  No prospective retina photographs but ongoing follow-up for reported changes in ARM status.
  A saliva or blood sample for genetic testing.
  Groups: ARM affected individuals and relatives.

SUMMARY:
The original study (GARM I) has been conducted for more than 18 years at the University of Pittsburgh Medical Center (UPMC). GARM II is a nationwide research study about age-related macular degeneration in the next generation of adults (49 to 65 years old). The purpose of this study is to identify the hereditary and exposure risk factors that lead to the development of ARM (Age related maculopathy).

Participants will communicate with the research staff through a protected and confidential website and use this website to complete a number of questionnaires during the course of the study (see below). For genetic analyses, the participants will mail in easily self-collected saliva samples in special containers. Eye photographs and eye health records are sent to the research center from local sources through the Internet. Individuals are not expected to come to UCLA in order to participate.

https://jseiclinres.jsei.ucla.edu/garm/

Participants will be expected to answer questionnaires or surveys about medical history, ocular history and visual symptoms, family history, smoking, dietary supplements and light exposure.

DETAILED DESCRIPTION:
Age-related macular degeneration (ARM) is a major cause of vision loss in the elderly. It is thought that smoking and diet may contribute to the risk of developing the condition but it is clear that heredity plays a major role. Variations in two genes, CFH and HTRA1/ARMS2, have been found to strongly contribute to the risk of developing ARM, but there are additional genes that influence a person's chances of having this condition and how they will progress to vision loss. We are investigating these genetic variations that contribute to ARM so that we can eventually understand the causes of this complex condition. We study the genetic variations (SNPs) that are shared among ARM-affected individuals within families as well as compare the frequencies of genetic variations in ARM-affected individuals with those in unaffected persons who are matched in age, gender, and exposures. We are conducting studies with the DNA from our previous cohort of research participants as well as developing a prospective study of high-risk family members and their spouses to evaluate genetic risks and presymptomatic retinal changes. Our long-term goals are to develop new preventive therapies that can slow or halt the development of this disease and to be able to provide these treatments to those who are at greatest risk before they experience vision-threatening changes.

The goal of this study (GARM II) is to determine how the combination of genetic, dietary, health and exposure factors such as light, diet, and smoking contributes to one's risk of developing this condition. This is not a treatment study and does not involve any preventive therapies or direct treatments of ARM. We aim to find some insights for future preventive strategies through a group of people who are at a higher than normal risk for developing ARM (because of their family history) and their partners who represent the risk in the general population. Because ARM is a complex disease and is affected by many factors, we also want to know how other medical conditions may be associated or not with this eye condition.

Participants will communicate with the research staff through a protected, HIPAA-compliant and confidential website and use this website to complete a number of questionnaires during the course of the study. For genetic analyses, the participants will mail in easily self-collected saliva samples in special containers. Eye photographs and eye health records are sent to the research center from local sources through the Internet. Individuals are not expected to come to UCLA in order to participate.

https://jseiclinres.jsei.ucla.edu/garm/

ELIGIBILITY:
Inclusion Criteria:

* Individuals should have an email account and access to the Internet in order to use the website for this study. Individuals who are unfamiliar or physically challenged with using computers may have another person assist them with reviewing messages, questions and entering information and making inquiries.
* ARM at-risk individuals between the ages of 49 to 65 years old who have at least one parent either deceased or alive with diagnosis of macular degeneration. This group includes the "third generation children" of our original GARM study.
* Individuals between the ages of 49 to 65 years old who are either a spouse or partner of an ARM at-risk adult (those individuals described above with a parent diagnosed with ARM).
* Individuals who have vision loss from ARM and a known family history of ARM (at least a brother, sister, or a parent). These individuals should have at least one at-risk child between the ages of 49 to 65 years old who is willing to participate in this study.

Exclusion Criteria:

* Inability to give informed consent. Adaptations will be provided to allow those who are unable to read because of vision loss to participate in the informed consent process.(Proxy)
* For the at risk individuals and their spouses/partners, they will be excluded if they do not have access and the ability to use a computer that is connected to the Internet.

Min Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nationwide study
Sampling Method: Non-Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2011-10-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The incidence and prevalence of retinal findings associated with early (and more advanced) age-related maculopathy in the study cohorts. | 5 years
  The primary outcome measure is the presence or absence of early retinal changes with age-related maculopathy in order to develop and test a model which combines genetic, environmental and dietary risk factors to predict which at risk individuals are most likely to develop signs of age-related maculopathy within the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gorin, MD, PhD, Principal Investigator — Jules Stein Eye Institute, UCLA
Locations (2):
- United States (2):
  - Jules Stein Eye Institute, Dept. of Ophthalmology David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Jakobsdottir J, Gorin MB, Conley YP, Ferrell RE, Weeks DE. Interpretation of genetic association studies: markers with replicated highly significant odds ratios may be poor classifiers. PLoS Genet. 2009 Feb;5(2):e1000337. doi: 10.1371/journal.pgen.1000337. Epub 2009 Feb 6. PMID 19197355
- [Background] Jakobsdottir J, Conley YP, Weeks DE, Ferrell RE, Gorin MB. C2 and CFB genes in age-related maculopathy and joint action with CFH and LOC387715 genes. PLoS One. 2008 May 21;3(5):e2199. doi: 10.1371/journal.pone.0002199. PMID 18493315
- [Background] Tikellis G, Sun C, Gorin MB, Klein R, Klein BE, Larsen EK, Siscovick DS, Hubbard LD, Wong TY. Apolipoprotein e gene and age-related maculopathy in older individuals: the cardiovascular health study. Arch Ophthalmol. 2007 Jan;125(1):68-73. doi: 10.1001/archopht.125.1.68. PMID 17210854
- [Background] Gorin MB. A clinician's view of the molecular genetics of age-related maculopathy. Arch Ophthalmol. 2007 Jan;125(1):21-9. doi: 10.1001/archopht.125.1.21. PMID 17210848
- [Background] Conley YP, Jakobsdottir J, Mah T, Weeks DE, Klein R, Kuller L, Ferrell RE, Gorin MB. CFH, ELOVL4, PLEKHA1 and LOC387715 genes and susceptibility to age-related maculopathy: AREDS and CHS cohorts and meta-analyses. Hum Mol Genet. 2006 Nov 1;15(21):3206-18. doi: 10.1093/hmg/ddl396. Epub 2006 Sep 25. PMID 17000705
- [Background] Jakobsdottir J, Conley YP, Weeks DE, Mah TS, Ferrell RE, Gorin MB. Susceptibility genes for age-related maculopathy on chromosome 10q26. Am J Hum Genet. 2005 Sep;77(3):389-407. doi: 10.1086/444437. Epub 2005 Jul 26. PMID 16080115
- [Background] Gorin MB. The coming of age for age-related macular degeneration genetics. Ophthalmic Genet. 2005 Jun;26(2):57-9. doi: 10.1080/13816810590969914. No abstract available. PMID 16020307
- [Background] Conley YP, Thalamuthu A, Jakobsdottir J, Weeks DE, Mah T, Ferrell RE, Gorin MB. Candidate gene analysis suggests a role for fatty acid biosynthesis and regulation of the complement system in the etiology of age-related maculopathy. Hum Mol Genet. 2005 Jul 15;14(14):1991-2002. doi: 10.1093/hmg/ddi204. Epub 2005 Jun 1. PMID 15930014
- [Background] Gorin MB. A new vision for age-related macular degeneration. Eur J Hum Genet. 2005 Jul;13(7):793-4. doi: 10.1038/sj.ejhg.5201431. No abstract available. PMID 15856069
- [Background] Weeks DE, Conley YP, Tsai HJ, Mah TS, Schmidt S, Postel EA, Agarwal A, Haines JL, Pericak-Vance MA, Rosenfeld PJ, Paul TO, Eller AW, Morse LS, Dailey JP, Ferrell RE, Gorin MB. Age-related maculopathy: a genomewide scan with continued evidence of susceptibility loci within the 1q31, 10q26, and 17q25 regions. Am J Hum Genet. 2004 Aug;75(2):174-89. doi: 10.1086/422476. Epub 2004 May 27. PMID 15168325
- [Background] Conley YP, Gorin MB. The genetics of age-related macular degeneration. Medsurg Nurs. 2003 Aug;12(4):238-41, 259. PMID 14515603
- [Background] Weeks DE, Conley YP, Tsai HJ, Mah TS, Rosenfeld PJ, Paul TO, Eller AW, Morse LS, Dailey JP, Ferrell RE, Gorin MB. Age-related maculopathy: an expanded genome-wide scan with evidence of susceptibility loci within the 1q31 and 17q25 regions. Am J Ophthalmol. 2001 Nov;132(5):682-92. doi: 10.1016/s0002-9394(01)01214-4. PMID 11704029